CLINICAL TRIAL: NCT00724893
Title: Pegetron® Redipen™ Prospective Optimal Weight-based Dosing Response Program
Brief Title: Efficacy of Pegetron® Redipen™ Treatment and Treatment Compliance of Patients With Chronic Hepatitis C in Canada (P04423)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04423; MK-4031-267 (Other: Merck Study Number)
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stage 1 Participants: Participants with CHC receiving PegIFN-2b using Redipen™ formulation (1.5 mcg/kg) once weekly and ribavirin capsules (800-1400 mg) daily according to routine medical practice at participating study sites.
  Interventions: Biological: PegIFN-2b; Drug: Ribavirin
- Stage 2 Participants: Participants with CHC Genotype 1 receiving PegIFN-2b using Redipen™ formulation (1.5 mcg/kg) once weekly and ribavirin capsules (800-1400 mg) daily according to routine medical practice at participating study sites.
  Interventions: Biological: PegIFN-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: PegIFN-2b — PegIFN-2b powder for solution adminstered subcutaneously using the newly approved Redipen. Dosing per approved labeling
  Other Names: Pegetron®; Pegylated interferon alfa-2b; PegIntron; SCH 054031
Drug: Ribavirin — Ribavirin capsules administered orally. Dosing in accordance with approved labelling.
  Other Names: SCH 018908

SUMMARY:
Treatment compliance is a key success factor in obtaining the full benefit of Pegetron (peginterferon alfa-2b [PegIFN-2b] plus ribavirin combination) therapy for patients. Treatment-naïve patients with chronic hepatitis C (CHC) in Canada to whom Pegetron Redipen was prescribed will receive Pegetron Redipen therapy in accordance with approved labeling. The study will assess the effect of the newly approved Pegetron Redipen on treatment compliance and its effect on sustained virologic response rates. Sustained virologic response is defined as negative hepatitis C virus ribonucleic acid (HCV-RNA) six months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve patients with chronic hepatitis C
* Adults (>18 years of age)
* Prescribed Pegetron Redipen
* Must meet all requirements for treatment with Pegetron Redipen
* Must be able to obtain reimbursement of medication through private or provincial coverage

Exclusion Criteria:

* Active hepatitis B virus (HBV) infection (hepatitis B surface antigen [HBsAg] positive)
* HIV antibody positive
* Post liver transplant patients
* Any other exclusion criteria as per the product Monograph

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve patients with chronic hepatitis C undergoing treatment with Pegetron Redipen at approximately 100 centers in Canada.
Sampling Method: Probability Sample
Enrollment: 2430 (Actual)
Dates: Start 2005-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Participants: Participants with chronic hepatitis C (CHC) receiving PegIFN-2b using Redipen™ formulation (1.5 mcg/kg) once weekly and ribavirin capsules (800-1400 mg) daily according to routine medical practice at participating study sites.
Period: Overall Study
Arm/Group | Stage 1 Participants | Stage 2 Participants
Started | 1302 | 1128
Completed | 938 | 670
Not Completed | 364 | 458
Not completed — Adverse Event | 76 | 142
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of virologic response | 94 | 202
Not completed — Reason not specified | 193 | 7
Not completed — Patient choice | 0 | 26
Not completed — Geographic reasons | 0 | 11
Not completed — Incarceration | 0 | 9
Not completed — Substance abuse | 0 | 3
Not completed — Financial reasons | 0 | 2
Not completed — Assigned shorter treatment | 0 | 2
Not completed — Lost to Follow-up | 0 | 52
Not completed — Unknown, missing data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Participants | Stage 2 Participants | Total
Number analyzed (Participants) | 1302 | 1128 | 2430
Age, Customized [Number; unit: Participants]
  <25 years | 23 | 12 | 35
  24 to < 40 years | 275 | 217 | 492
  40 to < 55 yeats | 783 | 671 | 1454
  >55 years | 221 | 228 | 449
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 432 | 346 | 778
  Male | 870 | 782 | 1652

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Viral Response at Any Evaluation Point (Stage 1)
Description: This is a measure of the number of participants achieving a viral response (negative hepatitis C virus ribonucleic acid [HCV-RNA]) at either of the follow-up evaluation time points (12 weeks [window 10-14 weeks] or ≥22 weeks after the end of treatment (EOT). Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants | 685

2. Primary Outcome: Number of Participants Achieving Viral Response at 12 Weeks After EOT (Stage 1)
Description: This is a measure of the number of participants achieving a viral response (negative HCV-RNA) at 12 weeks (window 10-14 weeks) after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 62 weeks
Population: All participants who took at least one dose of study medication (ITT population)
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
Participants | 660

3. Primary Outcome: Number of Participants Achieving Sustained Viral Response (SVR) (Stage 1)
Description: This is a measure of the number of participants who achieved SVR, defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT population)
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
Participants | 638

4. Primary Outcome: Number of Participants Achieving SVR (Stage 2)
Description: SVR was defined as HCV-RNA negative at six months after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants | 468

5. Secondary Outcome: Number of Participants Discontinued From Study Treatment Due to Adverse Events (Stage 1 and Stage 2)
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment
Time Frame: Up to 48 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants | Stage 2 Participants
Number analyzed (Participants) | 1302 | 1128
participants | 76 | 142

6. Secondary Outcome: Number of Participants Achieving Viral Response at Any Evaluation Point, Excluding Participants Who Discontinued Treatment Prior to Early Virologic Response (EVR) Evaluation (Stage 1)
Description: Viral response was defined as negative HCV-RNA. EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative at Treatment Week 12. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: Participants in the ITT population with EVR evaluation at Treatment Week 12
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1213
Participants | 685

7. Secondary Outcome: Number of Participants Achieving Viral Response at 12 Weeks After EOT, Excluding Participants Who Discontinued Prior to EVR Evaluation (Stage 1)
Description: as for outcome 6
Time Frame: Up to 62 weeks
Population: Participants in the ITT population with EVR evaluation at Treatment Week 12
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1213
Participants | 660

8. Secondary Outcome: Number of Participants Achieving SVR, Excluding Participants Who Discontinued Prior to EVR Evaluation (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative at Treatment Week 12. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: Participants in the ITT population with EVR evaluation at Treatment Week 12
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1213
Participants | 638

9. Secondary Outcome: The Number of Participants Achieving Viral Response at 12 Weeks After EOT, Excluding Participants Who Discontinued Prior to EVR Evaluation and Participants With Missing Data (Stage 1)
Description: Viral response was defined as negative HCV-RNA; evaluation was done 12 weeks (window 10-14 weeks) after EOT. EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative at Treatment Week 12. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 62 weeks
Population: Participants in the ITT population with EVR evaluation at Treatment Week 12 and no missing data
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1126
Participants | 679

10. Secondary Outcome: The Number of Participants Achieving SVR Excluding Participants Who Discontinued Prior to EVR Evaluation and Participants With Missing Data (Stage 1)
Description: as for outcome 8
Time Frame: Up to 72 weeks
Population: Participants in the ITT population with EVR evaluation at Treatment Week 12 and no missing data
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1037
participants | 612

11. Secondary Outcome: The Number of Participants Achieving Viral Response at 12 Weeks After EOT by Chronic HCV Genotype (Stage 1)
Description: Viral response was defined as negative HCV-RNA; evaluation was done 12 weeks (window 10-14 weeks) after EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 62 weeks
Population: All participants who took at least one dose of study medication (ITT population).
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
Participants
  Genotype 1 (n=757) | 308
  Genotype 2 (n=172) | 129
  Genotype 3 (n=348) | 215
  Genotype 4 (n=21) | 6
  Genotype 5 (n=0) | 0
  Genotype 6 (n=2) | 2
  Genotype unknown (n=2) | 0

12. Secondary Outcome: The Number of Participants Achieving Viral Response at 12 Weeks After EOT by Liver Fibrosis Stage (Stage 1)
Description: Viral response was defined as negative HCV-RNA; evaluation was done 12 weeks (window 10-14 weeks) after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 =significant liver damage, the liver becomes fibrotic [scarred] and connects with other scarred areas, and F4 = severe damage [cirrhosis] and liver no longer functions properly).
Time Frame: Up to 62 weeks
Population: All participants who took at least one dose of study medication (ITT population)
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
Participants
  F0 (n=59) | 34
  F1 (n=159) | 89
  F2 (n=216) | 95
  F3 (n=128) | 51
  F4 (n=111) | 40
  Fibrosis stage unknown (n=629) | 351

13. Secondary Outcome: Number of Participants Achieving SVR by Liver Fibrosis Stage (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 = significant liver damage, the liver is fibrotic [scarred] and connects with other scarred areas, and F4 = severe damage [cirrhosis] and liver no longer functions properly).
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  F0 (n=59) | 33
  F1 (n=159) | 85
  F2 (n=216) | 90
  F3 (n=128) | 49
  F4 (n=111) | 38
  Fibrosis stage unknown (n=629) | 343

14. Secondary Outcome: Number of Participants Achieving SVR by Chronic HCV Genotype (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks following EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  Genotype 1 (n=757) | 298
  Genotype 2 (n=172) | 126
  Genotype 3 (n=348) | 207
  Genotype 4 (n=21) | 5
  Genotype 5 (n=0) | 0
  Genotype 6 (n=2) | 2
  Genotype missing (n=2) | 0

15. Secondary Outcome: Number of Participants Achieving SVR by Viral Load (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no". Viral load categories were defined as High (≥100,000 Iu/mL) or Low (<100,000 Iu/mL).
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  Viral load high (n=836) | 353
  Viral load low (n=109) | 63
  Viral load missing (n=357) | 222

16. Secondary Outcome: Number of Participants Achieving SVR by Weight (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  40 to <50 kg (n=21) | 10
  50 to <64 kg (n=160) | 82
  64 to <75 kg (n=297) | 158
  75 to <85 kg (n=283) | 137
  >85 kg (n=541) | 251

17. Secondary Outcome: Number of Participants Achieving SVR by Chronic HCV Genotype + Liver Fibrosis Stage (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 =significant liver damage, the liver becomes fibrotic [scarred] and connects with other scarred areas, and F4 = severe damage [cirrhosis] and liver no longer functions properly). For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population); no participants had Genotype 5
Measure: Number; unit: participants
Groups:
- Stage F0: Participants with Fibrosis Stage F0
- Stage F1: Participants with Fibrosis Stage F1
- Stage F2: Participants with Fibrosis Stage F2
- Stage F3; Stage F4: Participants with Fibrosis Stage F4
- Unknown Stage: Participants with unknown Fibrosis Stage
Arm/Group | Stage F0 | Stage F1 | Stage F2 | Stage F3 | Stage F4 | Unknown Stage
Number analyzed (Participants) | 59 | 159 | 216 | 128 | 111 | 629
participants
  Genotype 1 (n=757) | 21 | 55 | 64 | 28 | 25 | 105
  Genotype 2 (n=172) | 4 | 17 | 13 | 9 | 2 | 81
  Genotype 3 (n=348) | 8 | 13 | 13 | 10 | 9 | 154
  Genotype 4 (n=21) | 0 | 0 | 0 | 0 | 2 | 3
  Genotype 6 (n=2) | 0 | 0 | 0 | 2 | 0 | 0
  Unknown Genotype (n=2) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Achieving SVR by Chronic HCV Genotype + Viral Load (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no". Viral load categories were defined as High (≥100,000 Iu/mL) or Low (<100,000 Iu/mL). For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population); no participants had Genotype 5
Measure: Number; unit: participants
Groups:
- Viral Load High; Viral Load Low: Participants with viral load xxxx
- Viral Load Missing: Participants with viral load missing
Arm/Group | Viral Load High | Viral Load Low | Viral Load Missing
Number analyzed (Participants) | 836 | 109 | 357
participants
  Genotype 1 (n=757) | 222 | 42 | 34
  Genotype 2 (n=172) | 53 | 4 | 69
  Genotype 3 (n=348) | 74 | 14 | 119
  Genotype 4 (n=21) | 2 | 3 | 0
  Genotype 6 (n=2) | 2 | 0 | 0
  Unknown Genotype (n=2) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants Achieving SVR by Weight + Chronic HCV Genotype (Stage 1)
Description: SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population); no participants had Genotype 5
Measure: Number; unit: participants
Groups:
- 40 to <50 kg: Participants with weight 40 to <50 kg
- 50 to <64 kg: Participants with weight 50 to <64 kg
- 64 to <75 kg: Participants with weight 64 to <75 kg
- 75 to <85 kg: Participants with weight 75 to <85 kg
- >85 kg: Participants with weight >85 kg
Arm/Group | 40 to <50 kg | 50 to <64 kg | 64 to <75 kg | 75 to <85 kg | >85 kg
Number analyzed (Participants) | 21 | 160 | 297 | 283 | 541
participants
  Genotype 1 (n=757) | 4 | 39 | 76 | 61 | 118
  Genotype 2 (n=172) | 5 | 11 | 26 | 26 | 58
  Genotype 3 (n=348) | 1 | 31 | 53 | 47 | 75
  Genotype 4 (n=21) | 0 | 0 | 2 | 3 | 0
  Genotype 6 (n=2) | 0 | 1 | 1 | 0 | 0
  Genotype unknown (n=2) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants Achieving EVR (Stage 1)
Description: EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative after 12 weeks of treatment. Participants with no viral response information were considered viral response "no".
Time Frame: From Week 10 to Week 14
Population: The EVR analysis population comprised participants with HCV Genotypes 1, 4, and 6 only, who took at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 780
participants | 473

21. Secondary Outcome: Number of Participants Achieving SVR by EVR Type (Stage 1)
Description: EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative after 12 weeks of treatment. SVR was defined as HCV-RNA negative at ≥22 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: The EVR analysis population comprised participants with HCV Genotypes 1, 4, 5, and 6 who took at least one dose of study medication. No participants had Genotype 5.
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 473
participants
  EVR by ≥2 log reduction from baseline (n=78) | 15
  EVR by HCV-RNA negative (n=389) | 253
  EVR missing (n=6) | 2

22. Secondary Outcome: Number of Participants Achieving SVR by Gender (Stage 1)
Description: as for outcome 16
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  Female (n=432) | 241
  Male (n=870) | 397

23. Secondary Outcome: Number of Participants Achieving SVR by Race (Stage 1)
Description: as for outcome 16
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  Asian (n=78) | 59
  Black (n=18) | 9
  Caucasian (N=1110) | 524
  Hispanic (n=11) | 4
  Other (n=85) | 42

24. Secondary Outcome: Number of Participants Achieving SVR by Human Immunodeficiency Virus (HIV) Status (Stage 1)
Description: as for outcome 16
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants
  HIV positive (n=11) | 3
  HIV negative (n=1075) | 543
  HIV status not done (n=216) | 92

25. Secondary Outcome: Number of Participants With End of Treatment (EOT) Response (Stage 1)
Description: EOT response was defined as HCV-RNA negative after 24 weeks of treatment in participants with HCV Genotype 2 or 3, and after 48 weeks of treatment in participants with Genotype 1, 4, 5, or 6. If there was no EOT information or if it was marked as "not done" then EOT was set to "no".
Time Frame: Up to 48 weeks
Population: All participants who took at least one dose of study medication (ITT Population); no participants had Genotype 5
Measure: Number; unit: participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
participants | 800

26. Secondary Outcome: Number of Participants With EOT Response by Chronic HCV Genotype (Stage 1)
Description: EOT response was defined as HCV-RNA negative after 24 weeks of treatment in participants with HCV-RNA Genotype 2 or 3, and after 48 weeks of treatment in participants with Genotype 1, 4, 5, or 6. If there was no EOT information or if it was marked as "not done" then EOT was set to "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population); no participants had Genotype 5
Measure: Number; unit: particpants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
particpants
  Genotype 1, 4, and 6 (N=780) | 405
  Genotype 2 and 3 (n=520) | 395
  Genotype missing (n=2) | 0

27. Secondary Outcome: Number of Participants With EVR by Selected Chronic HCV Genotypes (Stage 1)
Description: EVR was defined as either HCV-RNA detectable with a ≥2 log reduction from baseline or HCV-RNA negative at TW12. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Week 12
Population: The EVR analysis population comprised participants with HCV genotypes 1, 4, and 6 only, who took at least one dose of study medication; no participants had Genotype 5
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 780
Participants
  Genotype 1 (n=757) | 461
  Genotypes 1,4, and 6 (n=780) | 473

28. Secondary Outcome: Relapse Rate by HCV Genotype (Stage 1)
Description: The relapse rate was calculated with these parameters: EOT "yes", EVR evaluation valid, and ≥22 weeks of follow-up data. There were no imputations for EOT or SVR. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 48 weeks
Population: All participants who took at least one dose of study medication (ITT population) and had EOT "yes" and valid EVR evaluation ; no participants had Genotype 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 598
Percentage of Participants
  Genotype 1 (n=251) | 11.5
  Genotype 2 (n=123) | 3.2
  Genotype 3 (n=217) | 9.7
  Genotype 4 (n=5) | 40.0
  Genotype 6 (n=2) | 0

29. Secondary Outcome: Number of Participants Discontinued From Study Drug Due to Adverse Events by Chronic HCV Genotype (Stage 1)
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment. For this analysis participants were grouped by their HCV genotype (Types 1-6); a genotype is a classification based on the differences in the genetic material within the hepatitis virus. Knowing the HCV genotype helps with deciding what type and what duration of treatment will be needed because each genotype demonstrates a different response to treatment in infected individuals.
Time Frame: Up to 48 weeks
Population: All participants who took at least one dose of study medication (ITT population); no participants had Genotype 5
Measure: Number; unit: Participants
Arm/Group | Stage 1 Participants
Number analyzed (Participants) | 1302
Participants
  Genotypes 1, 4, and 6 (n=780) | 52
  Genotype 2 and 3 (n=520) | 24

30. Secondary Outcome: Number of Participants Achieving Rapid Virologic Response (RVR) (Stage 2)
Description: RVR was defined as undetectable HCV-RNA after 4 weeks of treatment (window of 2 to 6 weeks). Participants with no viral response information were considered viral response "no".
Time Frame: Week 4
Population: The RVR analysis population comprised 388 participants who took at least one dose of study medication and were evaluated for RVR
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants | 56

31. Secondary Outcome: Number of Participants Achieving EVR (Stage 2)
Description: EVR was defined as either HCV-RNA undetectable with a ≥2 log reduction in HCV-RNA from baseline or HCV-RNA undetectable after 12 weeks of treatment. Participants with no viral response information were considered viral response "no".
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants | 690

32. Secondary Outcome: Number of Participants Achieving RVR by Race (Stage 2)
Description: as for outcome 30
Time Frame: Week 4
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants
  Aboriginal peoples/Metis (n=10) | 0
  Asian (n=19) | 6
  Black (n=8) | 0
  Caucasian (n=343) | 47
  Hispanic (n=1) | 0
  Other (n=7) | 3

33. Secondary Outcome: Number of Participants Achieving EVR by Race (Stage 2)
Description: as for outcome 31
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Aboriginal peoples/Metis (n=13) | 6
  Asian (n=54) | 42
  Black (n=20) | 8
  Caucasian (n=1002) | 609
  Hispanic (n=4) | 4
  Other (n=35) | 21

34. Secondary Outcome: Number of Participants Achieving SVR by Race (Stage 2)
Description: as for outcome 4
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Aboriginal peoples/Metis (n=13) | 4
  Asians (n=54) | 37
  Black (n=20) | 5
  Caucasian (n=1002) | 407
  Hispanic (n=4) | 4
  Other (n=35) | 11

35. Secondary Outcome: Number of Participants Achieving RVR Who Achieved SVR (Stage 2)
Description: RVR was defined as undetectable HCV-RNA after four weeks of treatment. SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Week 4
Population: Participants who achieved RVR
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 56
participants | 35

36. Secondary Outcome: Number of Participants Achieving EVR Who Achieved SVR (Stage 2)
Description: EVR was defined as either HCV-RNA undetectable with a ≥2 log reduction in HCV-RNA from baseline or HCV-RNA undetectable after 12 weeks of treatment. SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Week 12
Population: All participants who took at least one dose of study medication and achieved EVR
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 690
participants | 399

37. Secondary Outcome: Number of Participants Achieving RVR by Liver Fibrosis Stage (Stage 2)
Description: RVR was defined as undetectable HCV-RNA after four weeks of treatment. SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 =significant liver damage, the liver becomes fibrotic [scarred] and connects with other scarred areas , and F4 = severe damage [cirrhosis] and liver no longer functions properly).
Time Frame: Week 4
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants
  F0 (n=28) | 4
  F1 (n=30) | 9
  F2 (n=49) | 8
  F3 (n=14) | 2
  F4 (n=27) | 1
  Could not be determined (n=206) | 29
  Other (n=34) | 3

38. Secondary Outcome: Number of Participants Achieving EVR by Liver Fibrosis Stage (Stage 2)
Description: EVR was defined as either HCV-RNA undetectable with a ≥2 log reduction in HCV-RNA from baseline or HCV-RNA undetectable after 12 weeks of treatment.SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 =significant liver damage, the liver becomes fibrotic [scarred] and connects with other scarred areas , and F4 = severe damage [cirrhosis] and liver no longer functions properly).
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  F0 (n=66) | 49
  F1 (n=144) | 95
  F2 (n=212) | 133
  F3 (99) | 62
  F4 (n=110) | 53
  Could not be determined (n=463) | 280
  Other (n=34) | 18

39. Secondary Outcome: Number of Participants Achieving SVR by Liver Fibrosis Score (Stage 2)
Description: SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". Liver fibrosis stage was measured with the METAVIR scoring system (F0=no fibrosis or liver damage, F1 = beginning of liver damage with some slight scarring, F2 = moderate liver damage, scarring advancing in liver and surrounding blood vessels, F3 =significant liver damage, the liver becomes fibrotic [scarred] and connects with other scarred areas , and F4 = severe damage [cirrhosis] and liver no longer functions properly).
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  F0 (n=66) | 36
  F1 (n=144) | 72
  F2 (n=212) | 94
  F3 (n=99) | 35
  F4 (n=110) | 35
  Could not be determined (n=463) | 187
  Other (n=34) | 9

40. Secondary Outcome: Number of Participants Achieving RVR by Weight (Stage 2)
Description: RVR was defined as undetectable HCV-RNA after 4 weeks of treatment. Participants with no viral response information were considered viral response "no".
Time Frame: Week 4
Population: The RVR analysis population comprises 388 participants who took at least one dose of study medication and were evaluated for RVR
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants
  40 to <50 kg (n=3) | 0
  50-<64 kg (n=40) | 8
  64 to <75 kg (n=83) | 9
  75 to <85 kg (n=86) | 11
  >=85 kg (n=169) | 27
  Weight unknown (n=7) | 1

41. Secondary Outcome: Number of Participants Achieving EVR by Weight (Stage 2)
Description: as for outcome 31
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  40 to <50 kg (n=16) | 9
  50 to <64 kg (n=127) | 87
  64 to <75 kg (n=250) | 164
  75 to <85 kg (n=238) | 143
  >=85 kg (n=490) | 283
  Weight unknown (n=7) | 4

42. Secondary Outcome: Number of Participants Achieving SVR by Weight (Stage 2)
Description: SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  40 to <50 kg (n=16) | 6
  50 to <64 (n=127) | 59
  64 to <75 kg (n=250) | 115
  75 to >85 kg (n=238) | 93
  >=85 kg (n=490) | 193
  Weight unknown (n=7) | 2

43. Secondary Outcome: Number of Participants Achieving RVR by Chronic HCV Genotype 1 Subtype (Stage 2)
Description: RVR was defined as undetectable HCV-RNA after 4 weeks of treatment. SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype subcategory (1a or 1b); subcategories are the result of a change in the genetic material in the viruses within the genotype.
Time Frame: Week 4
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants
  Genotype 1a (n=147) | 17
  Genotype 1b (n=56) | 9
  Genotype unknown (n=160) | 26
  Genotype mixed (n=11) | 1
  Could not be determined (n=14) | 3

44. Secondary Outcome: Number of Participants Achieving EVR by Chronic HCV Genotype 1 Subtype (Stage 2)
Description: EVR was defined as either HCV-RNA undetectable with a ≥2 log reduction in HCV-RNA from baseline or HCV-RNA undetectable after 12 weeks of treatment.SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype subcategory (1a or 1b); subcategories are the result of a change in the genetic material in the viruses within the genotype.
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Genotype 1a (n=176) | 106
  Genotype 1b (n=74) | 51
  Genotype unknown (n=850) | 518
  Genotype mixed (n=14) | 8
  Could not be determined (n=14) | 7

45. Secondary Outcome: Number of Participants Achieving SVR by Chronic HCV Genotype 1 Subtype (Stage 2)
Description: SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no". For this analysis participants were grouped by their HCV genotype subcategory (1a or 1b); subcategories are the result of a change in the genetic material in the viruses within the genotype.
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Genotype 1a (n=176) | 58
  Genotype 1b (n=74) | 37
  Genotype Unknown (n=850) | 364
  Genotype mixed (n=14) | 5
  Could not be determined (n=14) | 4

46. Secondary Outcome: Number of Participants Achieving RVR by Gender (Stage 2)
Description: as for outcome 40
Time Frame: Week 4
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 388
participants
  Female (n=122) | 19
  Male (n=266) | 37

47. Secondary Outcome: Number of Participants Achieving EVR by Gender (Stage 2)
Description: as for outcome 31
Time Frame: Week 12
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Female (n=346) | 227
  Male (n=782) | 463

48. Secondary Outcome: Number of Participants Achieving SVR by Gender (Stage 2)
Description: as for outcome 42
Time Frame: Up to 72 weeks
Population: All participants who took at least one dose of study medication (ITT Population)
Measure: Number; unit: participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 1128
participants
  Female (n=346) | 167
  Male (n=782) | 301

49. Secondary Outcome: Number of Participants Achieving RVR by HIV Status (Stage 2)
Description: as for outcome 30
Time Frame: Week 4
Population: This analysis was not done.
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 0

50. Secondary Outcome: Number of Participants Achieving EVR by HIV Status (Stage 2)
Description: as for outcome 31
Time Frame: Week 12
Population: This analysis was not done.
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 0

51. Secondary Outcome: Number of Participants Achieving SVR by HIV Status (Stage 2)
Description: SVR was defined as HCV-RNA negative at six months following EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: This analysis was not done.
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 0

52. Secondary Outcome: Percentage of Compliance for Participants Achieving SVR Based on Medication Adherence Questionnaire (MAQ) (Stage 2)
Description: Compliance was defined as participants taking ≥80% versus <80% of their doses; compliance ≥80% was derived from participants who answered "always" or "most of the time" to Questions 4 (How often do you stick to your medication schedule for your Ribavirin?) and 5 (How often do you stick to your medication schedule for your Redipen [peginterferon] injections?) of the 6-question compliance questionnaire. Percentages are based on the total number of participants within each compliance category. SVR was defined as HCV-RNA negative at 24 weeks after EOT. Participants with no viral response information were considered viral response "no".
Time Frame: Up to 72 weeks
Population: Participants who completed the MAQ questionnaire during the study and achieved SVR
Measure: Number; unit: percentage of participants
Arm/Group | Stage 2 Participants
Number analyzed (Participants) | 314
percentage of participants
  Compliance < 80% (n=10) | 40.0
  Compliance ≥80% (n=304) | 39.1

ADVERSE EVENTS:
Description: No adverse events were collected for this study.
Arm/Group | Stage 1 Participants | Stage 2 Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No